CLINICAL TRIAL: NCT06614868
Title: Minority Stress Counseling for LGBTQ+ Individuals
Acronym: MST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Nicholas C. Borgogna, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300013570; NBLAB1 (Other: UAB)
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Minority Stress
Keywords: Minority Stress; Acceptance and Commitment Therapy
MeSH Terms: interventions — Acceptance and Commitment Therapy; Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Experimental): Participants receiving acceptance and commitment therapy
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Treatment as usual (Active Comparator): Unstructured counseling intervention
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — Up to 16 session of unstructured counseling therapy informed by Acceptance and Commitment Therapy tradition.
  Arms: Treatment Group
Behavioral: Treatment as Usual (TAU) — Unstructured counseling
  Arms: Treatment as usual

SUMMARY:
Lesbian, gay, bisexual, transgender, and queer+ (LGBTQ+) individuals experience a breadth of mental health disparities. Reducing these disparities is an area of key psychological research. Minority stress is theorized to be an underlying source of the disparities (Meyer, 2003). Minority stress can be conceptualized as the internalized stigma that results from experiences of social marginalization. By reducing minority stress, it is hypothesized that generalized mental illness indicators might be reduced and indicators of wellbeing increased.

DETAILED DESCRIPTION:
Adult participants will respond to advertisements by emailing a research assistant.

A research assistant will then arrange for a pre-screening interview to ensure inclusion criteria are met.

A research assistant will review informed consent and receive a signed informed consent during the pre-screening.

Participants who are accepted into the study will then be offered up to 12 sessions of ACT or receive an unstructured treatment as usual counseling condition delivered by graduate students in the UAB medical/clinical psychology program under the supervision of Dr. Borgogna. These sessions will be 45 minutes each and delivered in Dr. Borgogna's lab. During the first sessions a survey battery will be administered on a lab secure computer administered via Qualtrics. It will be re-administered at session six, and during the last session.

The survey will include a broad base of demographic, mental health, and minority stress measures.

Participants will be assigned a random number that will link their survey responses across sessions. Identifying information will not be gathered as part of data collection.

ELIGIBILITY:
Inclusion Criteria:

* Must identify as non-heterosexual

Exclusion Criteria:

Suicide attempt within the past 12 months.

Current eating disorder.

Narcotics use within the past 3 months

Non-suicidal self-injury within the past 6 months.

Current/History of psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Depression | 12 weeks
  Patient Health Questionnaire-9
Anxiety | 12 Weeks
  Generalized Anxiety Disorder-7
Post Traumatic Stress | 12 Weeks
  Patient Checklist-5
Internalized Heterosexism | 12 Weeks
  Internalized Homophobia Scale
Discrimination | 12 Weeks
  Daily Heterosexist Questionnaire
Alcohol Problems | 16 Weeks
  Alcohol Use Disorders Identification Test

SECONDARY OUTCOMES:
Experiential Avoidance | 16 Weeks
  Experiential Avoidance Rating Scale
Affect | 16 Weeks
  Positive Negative Affect Schedule
Problematic Pornography Use | 12 Weeks
  Brief Pornography Screen

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
deidentified data will be shared upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
URL: https://www.uab.edu/cas/psychology/people/faculty/nicholas-c-borgogna